CLINICAL TRIAL: NCT04939571
Title: European Disease Registry on Retinopathy of Prematurity (ROP)
Acronym: EU-ROP
Status: Recruiting | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: EU-ROP
Record Dates: First submitted 2021-06-01; First posted 2021-06-25 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Retinopathy of Prematurity
Keywords: ROP; anti-VEGF; laser coagulation; epidemiology; non-interventional study
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Preterm born infants treated for ROP
  Interventions: Other: Registry of preterm born infants with treatment-requiring ROP

INTERVENTIONS:
Other: Registry of preterm born infants with treatment-requiring ROP — All prematurely born infants who develop treatment requiring ROP and are treated (independent of the kind of treatment modality) at a center that participates in the registry are eligible for database entry.

SUMMARY:
The EU-ROP registry is a European wide multicenter non-interventional observational registry study intended to run open-ended in as many countries as possible including infants treated for retinopathy of prematurity irrespective of the used treatment modality. The registry is strictly observational; only clinical routine data is collected, no study-specific examinations or interventions are to be performed.

The aim of the EU-ROP registry is to collect information on as many patients as possible treated for ROP in Europe. Both the number of study centers as well as the number of patients to be included into the registry are not limited.

The primary objective is to describe the typical clinical features of infants with severe ROP, variations in phenotype, and the clinical progression of the disease over time (natural history) in different European countries as well as to study treatment patterns, follow-up patterns, as well as long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ROP requiring treatment according to the respective national ROP screening and treatment guidelines

Exclusion Criteria:

* Denial or absence of consent for documentation and electronic storage of personal data by parents or legal guardians

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All infants Europe wide with ROP requiring treatment can be entered into the registry. The aim of the EU-ROP registry is to collect information on as many patients as possible treated for ROP in Europe. Both the number of study centers as well as the number of patients to be included into the registry are not limited.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2038-08 (Estimated); Study Completion 2039-08 (Estimated)

PRIMARY OUTCOMES:
Baseline data of preterm born infants who develop treatment-requiring retinopathy of prematurity | Birth to treatment of ROP, an average of 12 weeks
  Birth weight, gestational age, weight at treatment, comorbidities (e.g. sepsis, necrotizing enterocolitis)
Treatment parameters at initial treatment | An average of 12 weeks postnatal age
  Type of treatment
Treatment parameters at re-treatment | Through study completion, an average of 20 to 30 weeks postnatal age
  Type of treatment
ROP stage | Through follow-up after treatment, an average of 1 year postnatal age
  Stage of ROP at treatment and during follow-up

SECONDARY OUTCOMES:
Long-term ophthalmic development | Up to 18 years
  Ophthalmic development (e.g. orthoptic status, visual acuity)
Long-term neurologic development | Up to 18 years
  Neurological developmental (e.g. assessed by psychometric assessments)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Stahl, Professor, Principal Investigator — Department of Ophthalmology, University Medicine Greifswald
Locations (59):
- University Eye Hospital Salzburg, Salzburg, Austria
- Bulgaria (3):
  - University Hospital Saint George, Plovdiv
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - University Eye Hospital Alexandrovska, Sofia
- University Eye Hospital Tartu, Tartu, Estonia
- Hospital Rothschild, Paris, France
- Germany (26):
  - University Eye Hospital, Aachen
  - University Eye Hospital Helios, Berlin
  - University Eye Hospital Vivantes, Berlin
  - University Eye Hospital Bonn, Bonn
  - Braunschweig Muncipal Hospital, Braunschweig
  - University Eye Hospital, Chemnitz
  - University Eye Hospital, Cologne
  - Carl-Thiem University Hospital Cottbus, Cottbus
  - University Eye Hospital, Düsseldorf
  - University Eye Hospital, Freiburg im Breisgau
  - University Eye Hospital Fulda, Fulda
  - University Eye Hospital Gießen, Giessen
  - University Eye Hospital, Göttingen
  - University Eye Hospital, Greifswald
  - University Eye Hospital, Hamburg
  - University Eye Hospital Hannover, Hanover
  - Facharztpraxis für Augenheilkunde, Ludwigshafen
  - University Eye Hospital, Lübeck
  - Ludwig-Maximilins-University Munich, Munich
  - Augenzentrum am St. Franziskus-Hospital, Münster
  - University Eye Hospital, Münster
  - Nuremberg South Hospital, Nuremberg
  - Ernst-von-Bergmann Hospital, Potsdam
  - University Eye Hospital, Regensburg
  - University Eye Hospital, Tübingen
  - University Eye Hospital Ulm, Ulm
- Greece (3):
  - P&A Kyriakou Athens Children Hospital, Athens
  - Department of Ophthalmology University Hospital of Larissa, Larissa
  - Aristotle University of Thessaloniki, Thessaloniki
- University Clinical Center of Kosovo, Pristina, Kosovo
- Poland (6):
  - Medical University of Bialystok Children's Clinical Hospital, Bialystok
  - University Hospital in Bydgoszcz, Bydgoszcz
  - University Hospital in Zabrze Silesia, Katowice
  - Prof. Dr. Stanislaw Popowski Regional Specialized Children's Hospital, Olsztyn
  - University of Medical Sciences Poznan, Poznan
  - Children's Memorial Health Institute Warsaw, Warsaw
- Spain (2):
  - Biomédica de Málaga y Plataforma en Nanomedicina, Málaga
  - University and Polytechnic Hospital La Fe, Valencia
- University Eye Hospital Genève, Geneva, Switzerland
- Turkey (Türkiye) (11):
  - University Eye Hospital Cukurova, Adana
  - Etlik Zübeyde Hanim Women's Health Education and Research Hospital, Ankara
  - Hacettepe University Children's Hospital, Ankara
  - University Eye Hospital Ankara, Ankara
  - University Eye Hospital Baskent, Ankara
  - University Eye Hospital Gazi, Ankara
  - University Eye Hospital Uludag, Bursa
  - Umraniye Research and Education Hospital, Istanbul
  - University Eye Hospital Koc, Istanbul
  - Ordu University Medical Faculty, Ordu
  - Ondokuz Mayis University Eye Hospital, Samsun
- Ukraine (3):
  - Department of Pediatric Ophthalmology and Eye Microsurgery Perinatal Center Kiev, Kiev
  - Kyiv Pediatric Hospital Ohmatdyt, Kiev
  - Filatov Institute of Eye Diseases and Tissue Therapy Odessa, Odesa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catt C, Pfeil JM, Barthelmes D, Gole GA, Krohne TU, Wu WC, Kusaka S, Zhao P, Dai S, Elder J, Heckmann M, Stack J, Khonyongwa-Fernandez G, Stahl A. Development of a joint set of database parameters for the EU-ROP and Fight Childhood Blindness! ROP Registries. Br J Ophthalmol. 2024 Jun 20;108(7):1030-1037. doi: 10.1136/bjo-2023-323915. PMID 37704267
- [Result] Winter K, Pfeil JM, Engmann H, Aisenbrey S, Lorenz B, Hufendiek K, Breuss H, Khattab M, Susskind D, Kakkassery V, Lagreze WA, Barth T, Liegl R, Brunder MC, Skevas C, Goldammer I, Glitz B, Michalewicz E, Krohne TU, Bartmann IR, Stahl A; Retina.net ROP and EU-ROP registry study groups. Comparability of input parameters in the German Retina.net ROP registry and the EU-ROP registry - An exemplary comparison between 2011 and 2021. Acta Ophthalmol. 2024 May;102(3):e314-e321. doi: 10.1111/aos.15753. Epub 2023 Sep 19. PMID 37725047
- See also: Project website — http://www.eu-rop.org